CLINICAL TRIAL: NCT02185560
Title: Drug Use Investigation of Sorafenib/ NEXAVAR® for Unresectable Differentiated Thyroid Carcinoma (DTC)
Brief Title: Prospective, Non-interventional, Post-authorization Safety Study That Includes All Patients Diagnosed as Unresectable Differentiated Thyroid Carcinoma and Treated With Sorafenib
Acronym: JPMS-DTC
Status: Active, not recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 17391; NEXAVAR-TC-01 (Other: Company Internal)
Record Dates: First submitted 2014-07-04; First posted 2014-07-09 (Estimated); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Thyroid Carcinoma
Keywords: Sorafenib; Differentiated Thyroid Carcinoma,; Japan; Post Marketing Surveillance; Drug Use Investigation
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BAY43-9006: NEXAVAR treatment group
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Patients treated by Physician with Nexavar under approved local prescriptions

SUMMARY:
This is a non-interventional, multi center post-authorization safety study that includes all patients diagnosed as Unresectable Differentiated Thyroid Carcinoma (DTC) and treated with Sorafenib within a certain period. The investigator should have made the choice of treatment (NEXAVAR) according with the Japanese Package Insert prior to enrolling the patient in this study.

The enrollment period is of 9 months. The observation period for each patient starts when the therapy with NEXAVAR is initiated. Patients will be followed for 9 months or until it is no longer possible (e.g. lost to follow-up); this will be considered the standard observation period. Those patients, to whom a total of 24 month follow up is possible, information on effectiveness including treatment duration and survival status of the patient and of keratoacanthoma and/or squamous cell cancer development will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients who start NEXAVAR treatment for radioactive iodine-refractory unresectable Differentiated Thyroid Carcinoma (DTC)

Exclusion Criteria:

* Patients who have already received NEXAVAR treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with Sorafenib for Unresectable Differentiated Thyroid Carcinoma (DTC)
Sampling Method: Non-Probability Sample
Enrollment: 453 (Actual)
Dates: Start 2014-06-27 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse drug reaction as a measure of safety and tolerability. | Up to 9 months
Number of participants with Serious adverse events as a measure of safety and tolerability. | Up to 9 months
Number of participants with Serious adverse drug reaction as a measure of safety and tolerability | Up to 9 months

SECONDARY OUTCOMES:
2-year survival | At 24 months
  Percentage of participants who survived 2 years from start of treatment
Time of treatment failure (TTF) | Up to 24 months
  Time to treatment failure is defined as the time interval from start of Nexavar therapy to the date of permanent discontinuation for any reason including disease progression, adverse event, patient preference or death.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Japan

REFERENCES:
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — http://clinicaltrials.bayer.com/